CLINICAL TRIAL: NCT04219826
Title: A Multi-Center, Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CK-3773274 in Adults With Symptomatic Hypertrophic Cardiomyopathy
Brief Title: Dose-finding Study to Evaluate the Safety, Tolerability, PK, and PD of CK-3773274 in Adults With HCM
Acronym: REDWOOD-HCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CY 6021; 2019-002785-12 (EudraCT Number)
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2023-11

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: CK-3773274; CK-274; obstructive hypertrophic cardiomyopathy; oHCM; REDWOOD-HCM; non-obstructive hypertrophic cardiomyopathy; nHCM; hypertrophic cardiomyopathy; HCM; aficamten
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CK-3773274 - Cohort 1 (Obstructive HCM) (Experimental): Subjects will receive doses of 5 - 15 mg of CK-3773274 with dose levels guided by echocardiography assessments for up to 10 weeks
  Interventions: Drug: CK-3773274 (5 - 15 mg)
- Placebo - Cohort 1 (Obstructive HCM) (Placebo Comparator): Subjects will receive placebo for up to 10 weeks
  Interventions: Drug: Placebo for CK-3773274
- CK-3773274 - Cohort 2 (Obstructive HCM) (Experimental): Subjects will receive doses 10 - 30 mg of CK-3773274 with dose levels guided by echocardiography assessments for up to 10 weeks
  Interventions: Drug: CK-3773274 (10 - 30 mg)
- Placebo - Cohort 2 (Obstructive HCM) (Placebo Comparator): Subjects will receive placebo for up to 10 weeks
  Interventions: Drug: Placebo for CK-3773274
- CK-3773274 & disopyramide - Cohort 3 (Obstructive HCM) (Experimental): Subjects will receive doses 5 - 15 mg of CK-3773274 with dose levels guided by echocardiography assessments for up to 10 weeks while taking disopyramide
  Interventions: Drug: CK-3773274 (5 - 15 mg)
- CK-3773274 - Cohort 4 (non-obstructive HCM) (Experimental): Subjects will receive doses of 5 - 15 mg of CK-3773274 with dose levels guided by echocardiography assessments for up to 10 weeks
  Interventions: Drug: CK-3773274 (5 - 15 mg)

INTERVENTIONS:
Drug: CK-3773274 (5 - 15 mg) — CK-3773274 tablets administered orally
  Arms: CK-3773274 & disopyramide - Cohort 3 (Obstructive HCM); CK-3773274 - Cohort 1 (Obstructive HCM); CK-3773274 - Cohort 4 (non-obstructive HCM)
Drug: CK-3773274 (10 - 30 mg) — CK-3773274 tablets administered orally
  Arms: CK-3773274 - Cohort 2 (Obstructive HCM)
Drug: Placebo for CK-3773274 — Placebo administered orally
  Arms: Placebo - Cohort 1 (Obstructive HCM); Placebo - Cohort 2 (Obstructive HCM)

SUMMARY:
This study is being performed to understand the effect of different doses of CK-3773274 on patients with hypertrophic cardiomyopathy (HCM).

ELIGIBILITY:
Inclusion Criteria

* Males and females between 18 and 85 years of age at screening.
* Body weight is ≥45 kg at screening.
* Diagnosed with HCM per the following criteria:

  * Has left ventricular (LV) hypertrophy with non-dilated LV chamber in the absence of other cardiac disease.
  * Has minimal wall thickness ≥15 mm (minimal wall thickness ≥13 mm is acceptable with a positive family history of HCM or with a known disease-causing gene mutation).
* Adequate acoustic windows for echocardiography.
* For Cohorts 1, 2 and 3 has LVOT-G during screening as follows:

  * Resting gradient ≥50 mmHg OR
  * Resting gradient ≥30 mmHg and <50 mmHg with post-Valsalva LVOT-G ≥50 mmHg
* For Cohort 4 has resting and post-Valsalva LVOT-G < 30 mmHg at the time of screening
* For Cohort 4 has elevated NT-proBNP > 300 pg/mL at the time of screening
* LVEF ≥60% at screening.
* New York Heart Association (NYHA) Class II or III at screening.
* Patients on beta-blockers, verapamil, diltiazem, or ranolazine should have been on stable doses for >4 weeks prior to randomization and anticipate remaining on the same medication regimen during the study.
* For Cohort 3: Patients must be taking disopyramide. Patients should have been on stable disopyramide doses for >4 weeks prior to screening and anticipate remaining on the same medication regimen during the study.

Exclusion Criteria

* Aortic stenosis or fixed subaortic obstruction.
* Known infiltrative or storage disorder causing cardiac hypertrophy that mimics oHCM (eg, Noonan syndrome, Fabry disease, amyloidosis).
* History of LV systolic dysfunction (LVEF <45%) at any time during their clinical course.
* Documented history of current obstructive coronary artery disease (>70% stenosis in one or more epicardial coronary arteries) or documented history of myocardial infarction.
* Has been treated with septal reduction therapy (surgical myectomy or percutaneous alcohol septal ablation) or has plans for either treatment during the study period (Cohorts 1, 2, and 3 only). Patients having undergone septal reduction therapy > 12 months prior to screening who remain symptomatic from nHCM, and who meet all other criteria for inclusion, may be enrolled in Cohort 4.
* For Cohorts 1, 2 and 4: Has been treated with disopyramide or antiarrhythmic drugs that have negative inotropic activity within 4 weeks prior to screening. (For Cohort 3, use of disopyramide is required).
* Has any ECG abnormality considered by the investigator to pose a risk to patient safety (eg, second degree atrioventricular block type II).
* Paroxysmal atrial fibrillation or flutter documented during the screening period.
* Paroxysmal or permanent atrial fibrillation requiring rhythm restoring treatment (eg, direct-current cardioversion, ablation procedure, or antiarrhythmic therapy) ≤6 months prior to screening. (This exclusion does not apply if atrial fibrillation has been treated with anticoagulation and adequately rate-controlled for >6 months).
* History of syncope or sustained ventricular tachyarrhythmia with exercise within 6 months prior to screening.
* Has received prior treatment with CK-3773274 or mavacamten.
* For Cohort 4: has any documented history of LVOT-G ≥ 30 mmHg at rest, with Valsalva, or with exercise (for subjects who have had prior septal reduction therapy, this exclusion criteria only applies to gradients detected following septal reduction therapy).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events observed during dosing of CK--3773274 in patients with HCM | 14 weeks
  Patient incidence of reported adverse events (AEs)

SECONDARY OUTCOMES:
Incidence of left ventricular ejection fraction (LVEF) < 50% observed during dosing of CK-3773274 in patients with HCM | 14 weeks
  Patient incidence of left ventricular ejection fraction (LVEF) < 50%
Incidence of serious adverse events observed during dosing of CK-3773274 in patients with HCM | 14 weeks
  Patient incidence of reported serious adverse events (SAEs)
Concentration-response relationship of CK-3773274 on the resting left ventricular outflow tract gradient (LVOT-G) on echocardiogram over 10 weeks of treatment in patients with oHCM (Cohorts 1, 2, 3 only) | 10 weeks
  Slope of the relationship of the plasma concentration of CK-3773274 to the change from baseline in the resting LVOT-G
Concentration-response relationship of CK-3773274 on the post-Valsalva left ventricular outflow tract gradient (LVOT-G) on echocardiogram over 10 weeks of treatment in patients with oHCM (Cohorts 1, 2, 3 only) | 10 weeks
  Slope of the relationship of the plasma concentration of CK-3773274 to the change from baseline in the post-Valsalva LVOT-G
Dose response relationship on LVOT-G of CK-3773274 in patients with oHCM at rest (Cohorts 1, 2, 3 only) | 10 weeks
  Change from baseline in resting LVOT-G over time as a function of dose
Dose response relationship on LVOT-G of CK-3773274 in patients with oHCM post-Valsalva (Cohorts 1, 2, 3 only) | 10 weeks
  Change from baseline in post-Valsalva LVOT-G over time as a function of dose
Concentration-response relationship of CK-3773274 on left ventricular ejection fraction (LVEF) over 10 weeks of treatment in patients with HCM | Day 1 to End of Study (EOS) (Week 14)
  Change from baseline in the resting LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics, MD, Study Director — Cytokinetics
Locations (22):
- United States (18):
  - Cedar-Sinai Medical Center, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Northwestern University, Evanston, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Medicine - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New York University Langone Health Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Cardiology at Southpoint, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania (University of Pennsylvania School of Medicine), Philadelphia, Pennsylvania
  - UMPC Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy
- Erasmus University Medical Center (Erasmus MC), Rotterdam, Netherlands
- Spain (2):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masri A, Sherrid MV, Abraham TP, Choudhury L, Garcia-Pavia P, Kramer CM, Barriales-Villa R, Owens AT, Rader F, Nagueh SF, Olivotto I, Saberi S, Tower-Rader A, Wong TC, Coats CJ, Watkins H, Fifer MA, Solomon SD, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Meng L, Sohn RL, Wohltman A, Maron MS; REDWOOD-HCM Investigators. Efficacy and Safety of Aficamten in Symptomatic Nonobstructive Hypertrophic Cardiomyopathy: Results From the REDWOOD-HCM Trial, Cohort 4. J Card Fail. 2024 Nov;30(11):1439-1448. doi: 10.1016/j.cardfail.2024.02.020. Epub 2024 Mar 15. PMID 38493832
- [Derived] Zampieri M, Argiro A, Marchi A, Berteotti M, Targetti M, Fornaro A, Tomberli A, Stefano P, Marchionni N, Olivotto I. Mavacamten, a Novel Therapeutic Strategy for Obstructive Hypertrophic Cardiomyopathy. Curr Cardiol Rep. 2021 Jun 3;23(7):79. doi: 10.1007/s11886-021-01508-0. PMID 34081217